CLINICAL TRIAL: NCT04022109
Title: Screening of Gastric Cancer Via Breath Volatile Organic Compounds by Hybrid Sensing Approach
Acronym: VOGAS
Status: Recruiting | Type: Observational
Sponsor: University of Latvia (Other)
Collaborators: Technion, Israel Institute of Technology (Other); University of Ulm (Other); Uppsala University (Other); JLM Innovation GmbH (Unknown); Universitaet Innsbruck (Other); Hospital Universitario San Ignacio (Other); Universidad de Pamplona (Other); Pontificia Universidad Catolica de Chile (Other); AC Camargo Cancer Center (Other); National Cancer Institute of Ukraine (Other); VTT Technical Research Centre of Finland (Other)
Responsible Party: Principal Investigator, Marcis Leja, Director, Institute of Clinical and Preventive Medicine, University of Latvia
Other Study IDs: 824986; lzp-2018/2-0228 (Other Grant/Funding Number: Latvia Research Council); KC-L-2017/5 (Other Grant/Funding Number: Investment and Development Agency of Latvia)
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer; Atrophic Gastritis; Gastric Dysplasia; H.Pylori Infection
Keywords: Volatile organic compounds; Breath testing; Gastric cancer; Atrophic gastritis; Precancerous lesions; Screening; Nanosensor technology; GC-MS
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled air samples being stored in specific adsorbent media Plasma/serum samples for group stratification Biopsy samples from stomach for histological assessment and microbiota analysis Gastric content samples for GC-MS and microbiota analysis Faecal samples for occult blood testing and microbiota analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Gastric cancer patients undergoing surgery: Patients with histologically confirmed gastric cancer (adenocarcinoma) planned for surgical management
  Interventions: Device: Breath sampling for VOC detection; Procedure: Surgery material collection for VOC headspace analysis; Diagnostic Test: Upper endoscopy; Diagnostic Test: Microbiota testing
- Gastric cancer patients: Patients with histologically confirmed gastric cancer (adenocarcinoma)
  Interventions: Device: Breath sampling for VOC detection; Diagnostic Test: Upper endoscopy; Diagnostic Test: Microbiota testing
- Control group patients without gastric cancer: Patients without gastric malignant disease according to data obtained in upper endoscopy
  Interventions: Device: Breath sampling for VOC detection; Diagnostic Test: Upper endoscopy; Diagnostic Test: Microbiota testing
- Average risk population: Average risk population of both genders aged 40-64 at the time of inclusion lacking alarm symptoms for gastrointestinal cancer
  Interventions: Device: Breath sampling for VOC detection; Diagnostic Test: Upper endoscopy; Diagnostic Test: Microbiota testing
- Patients with dyspeptic symptoms: Patients with dyspeptic symptoms or other complains being referred for upper endoscopy (Chile)
  Interventions: Device: Breath sampling for VOC detection; Diagnostic Test: Upper endoscopy; Diagnostic Test: Microbiota testing

INTERVENTIONS:
Device: Breath sampling for VOC detection — Breath sampling will be performed by using a special sensor device and or GC-MS analysis (by collecting breath samples in adsorbent tubes). Pepsinogen testing will be used in a subgroup to identify serological increased risk for atrophy
  Other Names: Serum, plasma sampling for group description and stratification
Procedure: Surgery material collection for VOC headspace analysis — Only for gastric cancer patients undergoing surgery (Group 1)
  Groups: Gastric cancer patients undergoing surgery
Diagnostic Test: Upper endoscopy — Routine endoscopic evaluation with a standard biopsy work-up according to updated Sydney system. Additional gastric contents for GC-MS and microbiota analysis in a subgroup. Endoscopy will be used only according to the clinical indications (in Group 4 - according to the results of pepsinogen tests)
  Other Names: Histological and microbial evaluation of biopsy samples and gastric content
Diagnostic Test: Microbiota testing — Faecal and gastric contents and biopsy samples for microbiota testing

SUMMARY:
The study is aimed to determine the potential of volatile marker testing for gastric cancer screening.

The study will be addressing the role of confounding factors, including lifestyle factors, diet, smoking as well as addressing the potential role of microbiota in the composition of exhaled volatile markers.

DETAILED DESCRIPTION:
Patients with established disease (gastric cancer, precancerous lesions) as well as patients investigated for the lesions and having been documented lack of the lesions will be enrolled to the study at clinical sites in Europe (Latvia, Ukraine) and Latin America (Colombia, Chile, Brazil). In addition, group of persons from general population at average risk for developing the target disease and individuals being referred for upper endoscopy according to clinical indications will be also enrolled.

Testing of volatile markers will be conducted by one of two methods: 1) gas chromatography coupled to mass spectroscopy (GS-MS) and 2) sensor technology. Various sensors will be used and evaluated for the purpose.

The potential sources of volatile organic compounds (VOCs) in the breath will be addressed by studying VOC emission by using headspace analysis from cancer tissue, gastric contents, cancer cell cultures and H.pylori.

The potential role of gastric and faecal microbiota in the origin of VOCs in the breath will be addressed. Metabolome in the circulation will also get correlated to VOCs in the breath and with microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with verified gastric cancer (Group 1 & 2)
* Patients undergoing or having undergone upper endoscopy according to clinical indications (Group 3 & 5)
* Average-risk population group aged 40-64 at inclusion without alarm symptoms (Group 4)
* Motivation to participate in the study
* Physical status allowing volatile marker sampling and other procedures within the protocol
* Signed consent

Exclusion Criteria:

* Known other active cancer
* Ventilation problems, airway obstruction
* Unwillingness or inability to co-operate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cancer patient population will be recruited in the major specialized cancer centres in Europe (Latvia, Ukraine) and Latin America (Colombia, Chile, Brazil) Control group patients will be recruited in the major specialized endoscopy centres in Europe (Latvia, Ukraine) and Latin America (Colombia, Chile, Brazil), most frequently - the same institutions as for cancer patient recruitment General population group (40-64 years) will be predominantly recruited in Latvia from the general population Symptomatic patient validation cohort (Group 5) will be predominantly recruited in Chile from the endoscopy referrals
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Characteristic VOC pattern identification for gastric cancer detection | 2 years following initiation of patient recruitment
  The characteristic VOC pattern based on sensor analysis and its performance indicators will be detected
Specific chemistry identification in the exhaled breath | 2 years following initiation of patient recruitment
  Identification of specific chemistries (GC-MS analysis) originating from gastric cancer

SECONDARY OUTCOMES:
Characteristic VOC pattern identification for gastric precancerous lesion detection | 2.5 years following initiation of patient recruitment
  The characteristic VOC pattern based on sensor analysis and its performance indicators will be detected
Identification of the best-performing sensors | 3 years following initiation of patient recruitment
  Comparative analysis between the performance of different sensor performance in target disease identification
Gut microbiota analysis in relation to breath VOCs | 3 years following initiation of patient recruitment
  Analysis of the role of gastric and faecal microbiota in the origin of VOCs in the exhaled breath

OTHER OUTCOMES:
Confounding factor analysis | 3 years following initiation of patient recruitment
  The role of confounding factors will be addressed to address their role in VOC emission

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Haick, PhD, Principal Investigator — TECHNION, Israel Institute for Technology
Locations (5):
- A.C.Camargo Cancer Center, São Paulo, Brazil
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Centro Javeriano de Oncología, San Ignacio University Hospital, Bogotá, Colombia
- Institute of Clinical and Preventive Medicine, University of Latvia, Riga, Latvia
- National Cancer Institute of Ukraine, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mochalski P, Leja M, Gasenko E, Skapars R, Santare D, Sivins A, Aronsson DE, Ager C, Jaeschke C, Shani G, Mitrovics J, Mayhew CA, Haick H. Ex vivo emission of volatile organic compounds from gastric cancer and non-cancerous tissue. J Breath Res. 2018 Jul 30;12(4):046005. doi: 10.1088/1752-7163/aacbfb. PMID 29893713
- [Background] Krilaviciute A, Stock C, Leja M, Brenner H. Potential of non-invasive breath tests for preselecting individuals for invasive gastric cancer screening endoscopy. J Breath Res. 2018 Apr 4;12(3):036009. doi: 10.1088/1752-7163/aab5be. PMID 29528036
- [Background] Amal H, Leja M, Funka K, Skapars R, Sivins A, Ancans G, Liepniece-Karele I, Kikuste I, Lasina I, Haick H. Detection of precancerous gastric lesions and gastric cancer through exhaled breath. Gut. 2016 Mar;65(3):400-7. doi: 10.1136/gutjnl-2014-308536. Epub 2015 Apr 13. PMID 25869737
- [Background] Krilaviciute A, Heiss JA, Leja M, Kupcinskas J, Haick H, Brenner H. Detection of cancer through exhaled breath: a systematic review. Oncotarget. 2015 Nov 17;6(36):38643-57. doi: 10.18632/oncotarget.5938. PMID 26440312
- [Background] Leja M, You W, Camargo MC, Saito H. Implementation of gastric cancer screening - the global experience. Best Pract Res Clin Gastroenterol. 2014 Dec;28(6):1093-106. doi: 10.1016/j.bpg.2014.09.005. Epub 2014 Sep 28. PMID 25439074
- [Background] Leja M, Amal H, Lasina I, Skapars R, Sivins A, Ancans G, Tolmanis I, Vanags A, Kupcinskas J, Ramonaite R, Khatib S, Bdarneh S, Natour R, Ashkar A, Haick H. Analysis of the effects of microbiome-related confounding factors on the reproducibility of the volatolomic test. J Breath Res. 2016 Jun 24;10(3):037101. doi: 10.1088/1752-7155/10/3/037101. PMID 27341527
- See also: Horizon 2020 project VOGAS web-page — https://www.vogas.eu/